CLINICAL TRIAL: NCT00004871
Title: Phase I, Dose De-Escalation to Minimal Effective Pharmacologic Dose Trial of Sodium Phenylbutyrate (PB, NSC 657802) in Combination With 5-Azacytidine (5-AZA, NSC 102816) in Patients With Myelodysplastic Syndromes (MDS) and Acute Myeloid Leukemia (AML)
Brief Title: Azacitidine Plus Phenylbutyrate in Treating Patients With Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067531, J9950; U01CA070095 (NIH); R01CA067803 (NIH); P30CA006973 (NIH); JHOC-99072307; NCI-T99-0092; JHOC-J9950
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; refractory anemia; refractory anemia with ringed sideroblasts; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Acute; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Azacitidine; 4-phenylbutyric acid

INTERVENTIONS:
Drug: azacitidine
Drug: sodium phenylbutyrate

SUMMARY:
RATIONALE: Azacitidine plus phenylbutyrate may help leukemia cells develop into normal white blood cells.

PURPOSE: Phase I trial to study the effectiveness of combining azacitidine and phenylbutyrate in treating patients who have acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and toxicity of azacitidine in combination with phenylbutyrate in patients with recurrent, refractory, or untreated acute myeloid leukemia or myelodysplastic syndrome.
* Determine the minimal effective pharmacologic dose of azacitidine required to consistently inhibit DNA methyltransferase in this patient population.
* Obtain preliminary clinical and/or laboratory data suggesting potential therapeutic activity of this combination regimen in these patients.

OUTLINE: This is a dose deescalation study of azacitidine.

Patients receive azacitidine subcutaneously daily on days 1-5 and 29-33 followed by phenylbutyrate IV continuously on days 5-12 and 33-40. Treatment continues for at least 2 courses in the absence of disease progression. Patients with responsive disease may receive an additional 2 months of therapy.

Cohorts of 3-6 patients receive deescalating doses of azacitidine until the minimal effective pharmacologic dose (MEPD) is determined. The MEPD is defined as the dose above the dose at which more than 1 of 6 patients do not meet the target enzyme inhibition of greater than 90%.

Once the MEPD and toxicity have been established for a 5 day schedule, daily dose schedule of azacitidine is increased to 10, 14, and 21 days, followed by phenylbutyrate for 7 days. Courses are repeated every 28 days.

PROJECTED ACCRUAL: Approximately 32 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed myelodysplastic syndrome (MDS) indicating one of the following:

  * Refractory anemia (RA)
  * Primary refractory leukopenia or thrombocytopenia with MDS morphology
  * RA with excess blasts (RAEB)
  * RA with ringed sideroblasts (RARS)
  * Chronic myelomonocytic leukemia
  * RAEB in transformation
* RA or RARS must have at least one of the following:

  * Absolute neutrophil count less than 1,000/mm^3
  * Untransfused hemoglobin less than 8 g/dL
  * Platelet count less than 20,000/mm^3
  * Anemia
  * Thrombocytopenia requiring transfusion
  * High risk chromosomal abnormalities
* Any stage of MDS allowed including:

  * Previously untreated MDS
  * Refractory MDS allowed if failure to achieve remission following prior intensive chemotherapy of at least 1 month ago
* Relapsed, refractory, or untreated acute myeloid leukemia (AML) with the following:

  * WBC less than 30,000/mm^3
  * Stable for at least 2 weeks
  * Unlikely to require cytotoxic therapy during study
* Untreated AML with poor risk factors for response to standard therapy including:

  * Greater than 60 years old
  * AML occurs in setting of antecedent hematologic disorder
  * High risk chromosomes (e.g., abnormalities of chromosome 5 or 7 or complex cytogenetic abnormalities)
  * Medical conditions that preclude cytotoxic chemotherapy as primary therapy
* Refusal of cytotoxic chemotherapy allowed
* No clinical evidence of CNS leukostasis or CNS leukemia

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics
* Hemoglobin at least 8 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 2.0 mg/dL (unless due to hemolysis or Gilbert's disease)

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* No disseminated intravascular coagulation

Pulmonary:

* No pulmonary leukostasis

Other:

* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception 2 weeks prior, during and 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy including colony stimulating factors and recovered

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy and recovered

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy and recovered

Radiotherapy:

* At least 3 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Steven D. Gore, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States